CLINICAL TRIAL: NCT02448537
Title: A Phase II Multi-Strata Study of PM01183 as a Single Agent or in Combination With Conventional Chemotherapy in Metastatic and/or Unresectable Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); PharmaMar (Industry)
Responsible Party: Principal Investigator, Gregory Cote, MD PhD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-083
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Results first posted 2018-03-05 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Metastatic Sarcoma
Keywords: Metastatic Sarcoma; Unresectable Sarcoma; PM01183
MeSH Terms: conditions — Sarcoma | interventions — PM 01183; Doxorubicin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PM01183 and Doxorubicin (Experimental): Anthracycline-naïve patients will receive combination of PM01183 and Doxorubicin per cycle.
  * PM01183 predetermined dose daily via IV per cycle
  * Doxorubicin predetermined dose daily via IV per cycle
  Interventions: Drug: PM01183; Drug: Doxorubicin
- PM01183 and Gemcitabine (Experimental): Prior anthracycline exposure and without prior gemcitabine exposure
  * PM01183 predetermined dose given twice via IV per cycle
  * Gemcitabine predetermined dose given twice via IV per cycle
  Interventions: Drug: PM01183; Drug: Gemcitabine
- Single Agent PM01183 (Experimental): Patients who have received at least both prior anthracycline and prior gemcitabine
  -PM01183 predetermined dose once via IV per cycle
  Interventions: Drug: PM01183

INTERVENTIONS:
Drug: PM01183
  Other Names: lurbinectedin
Drug: Doxorubicin
  Other Names: Hydroxydaunomycin Hydrochloride; Adriamycin; Hydroxydoxorubicin Hydrochloride
  Arms: PM01183 and Doxorubicin
Drug: Gemcitabine
  Other Names: Gemzar
  Arms: PM01183 and Gemcitabine

SUMMARY:
This research study is investigating a drug called PM01183 alone and in combination with chemotherapy drugs called gemcitabine or doxorubicin as a possible treatment for metastatic or unresectable Sarcoma.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

PM01183 is a new drug that is believed to bind DNA cause double strands of DNA to break. This drug has been studied in previous research studies, and these suggest that it may slow or stop the growth of cancers. The FDA (the U.S. Food and Drug Administration) has not approved PM01183 as a treatment for any disease.

In this research study, the investigators are trying to assess the effects, good or bad, that PM01183, administered either alone or in combination with gemcitabine or doxorubicin has on metastatic or unresectable sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have pathologically confirmed soft-tissue sarcoma, which is metastatic or unresectable, sarcoma with no curative multimodality options
* Participants must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* No more than two prior lines of chemotherapy for metastatic sarcoma are allowed; Neo-adjuvant/adjuvant chemotherapy with definitive therapy (radiation, surgery or radiation and surgery) will not be counted as one of these prior lines of therapy.
* Age ≥ 18 and ≤ 75 years.
* Eastern Cooperative Oncology Group performance status ≤1 (see Appendix A)
* Life expectancy of greater than 3 months
* Participants must have normal organ and marrow function as defined below:

  * Hemoglobin ≥ 9 g/dl
  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 100,000/mcL
  * total bilirubin ≤ 1.5 X ULN
  * AST(SGOT)/ALT(SGPT) ≤3 X ULN (including patients with liver metastases)
  * creatinine ≤1.5 X ULN
  * CPK < 2.5 X ULN
  * Albumin ≥ 3 g/dl
* Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to receiving study agents.
* For patients in stratum A, an echocardiogram or multiple gated acquisition scan (MUGA) demonstrating left ventricular ejection fraction > 50% is required within 30 days prior to study drug administration.
* Participants must be willing and able to comply with the study scheduled visits, laboratory tests, and other procedures outlined in the protocol.
* Pre-menopausal women must have a negative pregnancy test before study entry. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for at least six weeks after treatment discontinuation. Acceptable methods of contraception include intrauterine device (IUD), oral contraceptive, subdermal implant, double barrier and/or complete abstinence (non-periodic).
* Washout period prior to Day 1 Cycle 1:

  * ≥ 3 weeks since last chemotherapy or therapeutic radiation therapy (RT)
  * ≥ 4 weeks or 3 half-lives since prior antibody-based therapy, whichever is shorter
  * ≥ 2 weeks since any oral anti-neoplastic or oral investigational agent
  * Resolution of treatment-related toxicity to ≤ grade 1; alopecia and cutaneous toxicity are allowed ≤ grade 2.
  * ≥1 week since palliative RT
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior exposure to PM01183
* Patients who have received trabectedin (Yondelis, ET-743) or participated in the phase III clinical study of trabectedin NCT01343277 previously will not be eligible.
* For stratum A, patients must not have received prior anthracycline-based therapy (prior treatment with non-anthracyclines is permitted).
* For stratum B patients must have received prior anthracycline-based therapy (or have a contraindication to receiving this treatment) and must not have received prior gemcitabine
* For stratum C, patients must have received prior anthracycline or gemcitabine-based therapy, or had a contraindication to either or both
* Prior radiation treatment of >45 Gy to the pelvis
* Previously untreated Ewing Sarcoma and rhabdomyosarcoma
* Non-soft tissue sarcomas, such as osteosarcoma and chondrosarcoma are excluded
* Participants who are receiving any other investigational agents.
* Active hepatopathy of any origin including active hepatitis B and hepatitis C
* Participants with known uncontrolled brain metastases will be excluded from this clinical.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PM01183 or trabectedin (Yondelis, ET-743).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, chronic indwelling drains, history of interstitial pneumonitis or pulmonary fibrosis or psychiatric illness/social situations that would limit compliance with study requirements.
* Actively breastfeeding women unless it is interrupted during treatment and at least 6 weeks after treatment discontinuation.
* Known myopathy or persistent CPK elevations >2.5 ULN in two different determinations performed one week apart.
* Immunocompromised patients, including those with HIV.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Cote, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Cote GM, Choy E, Chen T, Marino-Enriquez A, Morgan J, Merriam P, Thornton K, Wagner AJ, Nathenson MJ, Demetri G, George S. A phase II multi-strata study of lurbinectedin as a single agent or in combination with conventional chemotherapy in metastatic and/or unresectable sarcomas. Eur J Cancer. 2020 Feb;126:21-32. doi: 10.1016/j.ejca.2019.10.021. Epub 2019 Dec 31. PMID 31896519

RESULTS

PARTICIPANT FLOW:
Groups:
- PM01183 and Doxorubicin: Anthracycline-naïve patients will receive combination of PM01183 and Doxorubicin per cycle.
  * PM01183 predetermined dose daily via IV per cycle
  * Doxorubicin predetermined dose daily via IV per cycle
  PM01183
  Doxorubicin
- PM01183 and Gemcitabine: Prior anthracycline exposure and without prior gemcitabine exposure
  * PM01183 predetermined dose given twice via IV per cycle
  * Gemcitabine predetermined dose given twice via IV per cycle
  PM01183
  Gemcitabine
- Single Agent PM01183: Patients who have received at least both prior anthracycline and prior gemcitabine
  -PM01183 predetermined dose once via IV per cycle
  PM01183
Period: Overall Study
Arm/Group | PM01183 and Doxorubicin | PM01183 and Gemcitabine | Single Agent PM01183
Started | 20 | 10 | 12
Completed | 19 | 9 | 11
Not Completed | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PM01183 and Doxorubicin | PM01183 and Gemcitabine | Single Agent PM01183 | Total
Number analyzed (Participants) | 20 | 10 | 12 | 42
Age, Continuous [Median (Full Range); unit: years] | 52.6 [31.8 to 74.2] | 44.2 [29.6 to 74.5] | 55.3 [30.0 to 71.7] | 51.9 [29.6 to 74.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 7 | 26
  Male | 7 | 4 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 18 | 8 | 11 | 37
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15 | 7 | 11 | 33
  Black or African-American | 2 | 1 | 0 | 3
  Asian | 1 | 0 | 0 | 1
  More Than One Race | 2 | 1 | 0 | 3
  Other | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 12 | 42

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate
Description: The number of participants that achieved either Stable Disease (SD) or a Partial Response (PR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) at 24 weeks.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 24 Weeks
Population: Two participants (one from the PM01183 and Doxorubicin arm and one from the PM01183 alone arm) were not able to be evaluated for response.
Measure: Count of Participants; unit: Participants
Arm/Group | PM01183 and Doxorubicin | PM01183 and Gemcitabine | Single Agent PM01183
Number analyzed (Participants) | 20 | 10 | 12
Participants | 13 | 2 | 3

2. Secondary Outcome: Overall Response Rate
Description: The overall response rate is the number of participants that achieved either Stable Disease (SD), a Partial Response (PR), or a Complete Response (CR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST v1.1). The overall response rate is the best response recorded from the start of treatment until disease progression/recurrence.
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Every 6 weeks for the first 8 cycles (cycle is 21 days) and then every 9 weeks thereafter until disease progression
Measure: Count of Participants; unit: Participants
Arm/Group | PM01183 and Doxorubicin | PM01183 and Gemcitabine | Single Agent PM01183
Number analyzed (Participants) | 20 | 10 | 12
Participants
  Complete Response | 0 | 0 | 0
  Partial Response | 7 | 1 | 0
  Stable Disease | 6 | 1 | 3
  Unknown | 1 | 0 | 1

3. Secondary Outcome: Treatment Related Serious Adverse Events
Description: Summary of the serious adverse events (SAE) experienced by participants that were deemed to be at least possibly related to PM01183 when administered alone or with Doxorubicin or Gemcitabine. Adverse events were assessed using Common Terminology Criteria for Adverse Events (CTCAE v4).
Time Frame: From the start of treatment until 30 days after the end of treatment
Measure: Number; unit: participants
Arm/Group | PM01183 and Doxorubicin | PM01183 and Gemcitabine | Single Agent PM01183
Number analyzed (Participants) | 20 | 10 | 12
participants
  Diarrhea | 1 | 0 | 1
  Febrile neutropenia | 1 | 1 | 0
  Lymphocyte count decreased | 2 | 1 | 0
  Nausea | 1 | 0 | 1
  Neutrophil count decreased | 4 | 4 | 1
  Platelet count decreased | 1 | 1 | 0
  Port Infection | 0 | 1 | 0
  Vomiting | 1 | 0 | 1
  White blood cell decreased | 3 | 1 | 0
  Any Treatment Related SAE | 4 | 5 | 2

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the end of treatment.Treatment continued until the participant had disease progression, intercurrent illness that prevented further administration of treatment, an unacceptable adverse event, the participant withdrew from the study, or until the treating investigator decided it would be in the participants best interest.
Groups:
- Stratum A: Anthracycline-naïve patients will receive combination of PM01183 and Doxorubicin per cycle.
  * PM01183 predetermined dose daily via IV per cycle
  * Doxorubicin predetermined dose daily via IV per cycle
  PM01183
  Doxorubicin
- Stratum B: Prior anthracycline exposure and without prior gemcitabine exposure
  * PM01183 predetermined dose given twice via IV per cycle
  * Gemcitabine predetermined dose given twice via IV per cycle
  PM01183
  Gemcitabine
- Stratum C: Patients who have received at least both prior anthracycline and prior gemcitabine
  -PM01183 predetermined dose once via IV per cycle
  PM01183
Arm/Group | Stratum A | Stratum B | Stratum C
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 6/20 | 6/10 | 4/12
Other Adverse Events (participants affected / at risk) | 20/20 | 10/10 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum A (N=20) | Stratum B (N=10) | Stratum C (N=12)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Infections and infestations - Other, Port Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, Spontaneous Bacterial Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (6) | 4 (5) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (6) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, Grade 3 Decompression and Spinal Stabilization (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 3 (5) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum A (N=20) | Stratum B (N=10) | Stratum C (N=12)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (9) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 9 (12) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 6 (6) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 2 (3) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Carbon monoxide diffusing capacity decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Cardiac disorders - Other, Heart Murmur (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, Systolic Ejection Murmur (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorders - Other, tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac disorders - Other, Unspecified (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (19) | 5 (6) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 6 (8) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 1 (1)
Ear and labyrinth disorders - Other, Ear Rash (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 3 (3) | 0 (0) | 1 (1)
Endocrine disorders - Other, Polydispia/Polyuria (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Esophageal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, Left Eyelid Stye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, Vision Straining (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 18 (28) | 8 (11) | 5 (5)
Fever (General disorders) | 1 (1) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Abdominal Cramps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Abdominal Pressure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Early Satiety (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Gas Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Intermittent Dysgeusia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Partial Small Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Abdominal Tenderness (General disorders) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Chest Aching (General disorders) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Duodenitis (General disorders) | 0 (0) | 1 (2) | 0 (0)
General disorders and administration site conditions - Other, Itchy Eyes (General disorders) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, Sensitivity to Smells (General disorders) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Shingles (General disorders) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Shoulder Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Transfusion Reaction (General disorders) | 0 (0) | 1 (3) | 0 (0)
General disorders and administration site conditions - Other, Vascular Rash (General disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 2 (2) | 2 (2)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 4 (4) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Immune system disorders - Other, Cold Sore (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, Left Great Toe, Mild, Localized (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Thrush (Immune system disorders) | 3 (3) | 0 (0) | 2 (2)
Infections and infestations - Other, unspecified (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 3 (3) | 1 (1)
Investigations - Other, Leg Swelling (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 1 (4)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 5 (8) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Intermittent Bodyaching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Toe Cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (25) | 5 (7) | 5 (6)
Nervous system disorders - Other, Light-Headedness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 3 (4) | 2 (3)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (4) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (6) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Renal and urinary disorders - Other, Cloudy Urine (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, Intermittent Urinary Pressure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, Urinary Hesitancy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin/subcutaneous tissue disorders; Other, Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin/subcutaneous tissue disorders; Other, Nail Change - Brittle (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin/subcutaneous tissue disorders; Other, Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin/subcutaneous tissue disorders; Other, Vascular Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (10) | 1 (1) | 3 (3)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 6 (6) | 2 (2) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 2 (2) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT02448537/Prot_SAP_000.pdf